CLINICAL TRIAL: NCT02865499
Title: Acarbose as a Safe Effective Modulator of Aging Deficits in Geriatric Subjects
Brief Title: Acarbose Anti-aging Effects in Geriatric Subjects (Substudy B & C)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Dean L. Kellogg, Jr, Professor, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSC20120304
Record Dates: First submitted 2016-06-17; First posted 2016-08-12 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-02

CONDITIONS: Aging
MeSH Terms: interventions — Acarbose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- acarbose (Experimental): all participants will receive acarbose
  Interventions: Drug: acarbose

INTERVENTIONS:
Drug: acarbose — acarbose treatment with meals

SUMMARY:
This study addresses a "lifespan approach to healthy development and aging" with direct relevance to humans by testing the anti-aging effects of acarbose in humans. It is a pilot study to: i) better estimate power for a larger trial, ii) establish the safety and potential beneficial effects of acarbose in non-diabetic elderly humans, and iii) determine whether the effects of acarbose on the microbiome likely play a role in its enhancement of longevity and/or healthy aging. These are essential initial steps for translating acarbose into an anti-aging human therapy.

DETAILED DESCRIPTION:
Treatment with acarbose, an α-glucosidase inhibitor, extends median lifespan by 22% in male mice. Acarbose is FDA-approved for use in humans and has been extensively employed for the management of diabetics; there have been few associated side effects reported. Acarbose is considered a very safe treatment. Thus, the investigators hypothesize that acarbose treatment could be used in elderly humans to elicit improvement in systems known to be negatively affected by aging. Since the outcomes of acarbose treatment may be differentially affected by age, it is imperative to test the drug directly in older subjects for its safety and efficacy. Towards this end, the investigators propose to perform a small pilot study assessing the effects of acarbose in ten elderly subjects, aged 75-95 years old. Briefly, a cohort of non-diabetics will be recruited; subjects will be in generally good health with all chronic diseases (hypertension, coronary artery disease, etc.) clinically stable. Trial participants will be studied before drug initiation (pre-treatment), during 3 months of acarbose (blood draws at 1 month and 3 months of treatment), and following termination of the drug (1 and 3 months post treatment) such that each subject will serve as his own control. Gut microbiome composition will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* age 70-95
* participants will be in good health with all chronic diseases (hypertension, coronary artery disease, etc.) clinically stable.
* participants must have adequate cognitive function to be able to give informed consent. This will be established by enrolling participants with CLOX 1 scores of ≥10.

Exclusion Criteria:

* unstable ischemic heart disease
* clinically significant pulmonary disease
* history of immunodeficiency or receiving immunosuppressive therapy
* history of a coagulopathy or receiving a medical condition requiring anticoagulation
* an estimated glomerular filtration rate of <30ml/min
* uncontrolled hypercholesteremia >350mg/dl;
* uncontrolled hypertriglyceridemia >500mg/dl
* diabetes
* history of skin ulcers or poor wound healing
* smoking
* liver disease treatment with drugs known to affect cytochrome P450 3A (diltiazem, erythromycin)

Ages: 70 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-06; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean L Kellogg, Jr, MD, PhD, Principal Investigator — University of Texas
Locations (1):
- UTHSCSA, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | Acarbose
Started | 8
Completed | 6
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Period: 8 Weeks
Arm/Group | Acarbose
Started | 6
Completed | 6
Not Completed | 0
Period: 12 Weeks
Arm/Group | Acarbose
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Acarbose: all participants to receive acarbose
  acarbose: acarbose treatment with meals
Arm/Group | Acarbose
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Microbiome
Description: Changes in bacterial community measurement through DNA extraction from stool samples. Change is measured using operational taxonomic units (OTU). An OTU is the group of organisms being studied through DNA to cluster sequences of microbiomes according to their similarity to one another (the similarity threshold is set to 97%). This outcome measures change in the number of OTUs from baseline to 12 weeks.
Time Frame: Baseline; 8 weeks and 12 weeks
Measure: Number; unit: Operational Taxonomic Unit (OTU)
Groups:
- Acarbose: Stool specimens from all participants analyzed after acarbose
Arm/Group | Acarbose
Number analyzed (Participants) | 6
Operational Taxonomic Unit (OTU)
  Baseline Measurement | 0
  8 Week Measurement | 0
  12 Week Measurment | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Acarbose
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Budgetary restraints

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT02865499/Prot_SAP_000.pdf